CLINICAL TRIAL: NCT02907164
Title: Using Social Norms to Encourage People to Exercise More
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Hengchen Dai, Assistant Professor of Organizational Behavior, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201608038
Record Dates: First submitted 2016-09-03; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Group 1: Control (Active Comparator): People receive emails encouraging them to sign up for the challenge. The email does not mention the number of people who have signed up.
  Interventions: Behavioral: Email invitation
- Group 2: Norm (Experimental): People receive emails encouraging them to sign up for the challenge. The email mentions the number of people who have signed up.
  Interventions: Behavioral: Email invitation; Behavioral: Social norm
- Group 3: Norm and health motive (Experimental): People receive emails encouraging them to sign up for the challenge. The email mentions the number of people who have signed up AND highlights that the challenge helps people to stay fit in a fun way.
  Interventions: Behavioral: Email invitation; Behavioral: Social norm; Behavioral: Intrinsic, health motive
- Group 4: Norm and reward motive (Experimental): People receive emails encouraging them to sign up for the challenge. The email mentions the number of people who have signed up AND highlights that the challenge helps people to stay active and earn rewards.
  Interventions: Behavioral: Email invitation; Behavioral: Social norm; Behavioral: Extrinsic, reward motive

INTERVENTIONS:
Behavioral: Email invitation — Receive emails encouraging them to sign up
Behavioral: Social norm — Receive information about how many people have signed up
  Arms: Group 2: Norm; Group 3: Norm and health motive; Group 4: Norm and reward motive
Behavioral: Intrinsic, health motive — Receive information about how the challenge helps people to stay fit in a fun way
  Arms: Group 3: Norm and health motive
Behavioral: Extrinsic, reward motive — Receive information about how the challenge helps people to stay active and earn rewards
  Arms: Group 4: Norm and reward motive

SUMMARY:
The investigators are interested in using social norms to motivate people to sign up for a 100-day exercise challenge and exploring how to make social norms messages more effective.

DETAILED DESCRIPTION:
The investigators are interested in using social norms to motivate people to sign up for a 100-day exercise challenge and exploring how to make social norms messages more effective. Specifically, the primary purposes of this study are to test (a) whether social norms messages (i.e., information about how many people have signed up for the challenge) can increase signup rates and eventually lead people to exercise more and (b) whether such messages become more effective when they highlight different types of motivations (intrinsic vs. extrinsic motivations). Through a partnership with a university, the investigators are running a large-scale, randomized field controlled trial aimed at increasing sign-ups for the challenge and exercise frequencies during the challenge.

Benefits-eligible employees at the partner university are randomly assigned to one of four experimental conditions and receive the corresponding version of email message encouraging them to sign up for the challenge.

(1) In the control group, the email does not mention the number of people who have signed up. (2) In the norm condition, the email mentions the number of people who have signed up. (3) In the norm and health motive condition, the email mentions the number of people who have signed up, and highlights that the challenge is designed to help people to stay fit in a fun way. (4) In the norm and reward motive condition, the email mentions the number of people who have signed up, and highlights that the challenge is designed to help people to stay active and earn rewards.

The investigators hypothesize that Groups 2, 3, and 4 will have a higher sign-up rate and higher exercise frequencies on average than Group 1, because positive social norms should motivate people to engage in the target, desirable behavior. Also, the investigators will compare sign-up rates and exercise frequencies between Groups 2, 3, and 4 to examine whether highlighting intrinsic and extrinsic motives can further increase sign-up rates and overall exercise frequencies than only giving social norms information.

All benefits-eligible employees at the partner university for whom the Human Resource (HR) office has an email address on record receive invitation emails from HR. The invitation emails that contain the interventions are sent out one week AFTER the registration period has started, because HR needs to know how many people sign up in the first week and use this information to create a social norms message. Employees who sign up for the challenge during the first week of the registration period (i.e., prior to the implementation of the interventions) cannot be affected by the interventions. Thus, the investigators decide in advance that these employees will be excluded from analysis.

Employees will receive two emails that are sent eight days apart from each other. Thus, the investigators plan to examine both the sign-up rates within one week after each email goes out and the overall sign-up rates throughout the 50-day registration period.

The investigators plan to explore moderators based on (a) employees' demographics (age, gender, ethnicity, position), (b) employees' participation in previous challenges, and (c) employees' health condition and fitness level prior to the challenge (such as how actively they have been participating in other wellness activities, their health statistics).

ELIGIBILITY:
Inclusion Criteria:

* All benefits-eligible employees at partner university for whom the Human Resource office has an email address on record

Exclusion Criteria:

* Employees who sign up for the challenge prior to the implementation of the interventions will NOT be included in the analysis.

(The interventions are implemented one week after the registration period has started. The partner university has to send invitation emails to all benefits-eligible employees with an email address on record, including those who already signed up. However, employees who already signed up cannot be affected by the interventions and thus will be excluded from the analysis.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of people who sign up for the challenge | During the registration period, 50 days
  Whether or not each person signs up for the challenge during the registration period
Activity level | Through study completion, 100 days
  Number of steps taken each day, as recorded in participants' online portal

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Most recent BMI as entered by participant, an expected average of 2 months after study start
  most recent BMI in pounds (weight) and inches (height) as entered by participant, an expected average of 2 months after study start. Obtaining the data is dependent on the ability to obtain the data from the online portal.
cholesterol | Most recent cholesterol as entered by participant, an expected average of 2 months after study start
  Most recent total, low, and high cholesterol levels in mg/dl as entered by participant, an expected average of 2 months after study start. Obtaining the data is dependent on the ability to obtain the data from the online portal.
blood pressure | Most recent blood pressure as entered by participant, an expected average of 2 months after study start
  Most recent systolic and diastolic levels in mmHg as entered by participant, an expected average of 2 months after study start. Obtaining the data is dependent on the ability to obtain the data from the online portal.
stress | Most recent stress as entered by participant, an expected average of 2 months after study start
  Most recent self-reported stress level on a 1-5 scale (with 1 indicating "Relaxed" and 5 indicating "Highly Stressed") as entered by participant, an expected average of 2 months after study start. Obtaining the data is dependent on the ability to obtain the data from the online portal.
Email open and click rates | Through study completion, 100 days
  The rates at which people in each experimental condition read the invitation emails and click on links in the emails

CONTACTS AND LOCATIONS:
Overall Officials: Hengchen Dai, Ph.D, Principal Investigator — Washington University School of Medicine
Locations (1):
- Hengchen Dai, St Louis, Missouri, United States